CLINICAL TRIAL: NCT02322450
Title: Multicenter, Randomized, Double-blind, Two-period, Placebo Controlled, Forced-titration Proof of Concept Crossover Study to Compare QGC001 With Placebo in Patients With Grade I or II Essential Hypertension
Brief Title: Phase IIa Study of the Product QGC001 Compared With Placebo in Patients With Essential Hypertension
Acronym: 2QG1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quantum Genomics SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: QGC001/2QG1
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: P1-QGC001 - Washout-placebo - P2-placebo (Experimental): The first period (P1) will correspond either to QGC001 or placebo, the second period (P2) will correspond either to QGC001 or placebo.
  Interventions: Drug: QGC001; Drug: Placebo
- B: P1-placebo - Washout-placebo - P2-QGC001 (Experimental): The first period (P1) will correspond either to QGC001 or placebo, the second period (P2) will correspond either to QGC001 or placebo.
  Interventions: Drug: QGC001; Drug: Placebo

INTERVENTIONS:
Drug: QGC001
Drug: Placebo

SUMMARY:
2QG1 is a Phase IIa study aiming to assess the blood pressure lowering effect of 4-week administration of QGC001 oral doses in patients with grade I or II essential hypertension compared to placebo, to assess the safety and tolerability, to obtain preliminary PK information for QGC001 given as multiple oral doses and to determine preliminary PD profile of QGC001 multiple oral doses on plasma and urine hormones, which will be compared to that of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female of non-childbearing potential patients (post-menopausal since at least 12 months or surgically sterilized) aged 18 to 75 years;
* Body weight ≥50 kg with a body mass index (BMI) calculated as weight in kg/(height in m2) from 18 to 40 kg/m2 at screening;
* A signed and dated informed consent form before any study-specific screening procedure is performed;
* With a diagnosis of essential grade I or II hypertension defined as:

  * a supine office systolic BP (SBP) of 140-159 mmHg or diastolic BP (DBP) of 90-99 mmHg who should have an additional clinical indication according to ESH guidelines for antihypertensive treatment after a 2-week placebo run-in period,
  * or a supine office SBP of 160-179 mmHg or DBP of 100-109 mmHg after a 2-week placebo run-in period with a diagnosis of essential grade II hypertension;
* Diagnosis of permanent hypertension confirmed by a mean SBP or DBP higher than135 or 85 mmHg on daytime ambulatory blood pressure monitoring (ABPM) after a 2-week placebo run-in period;
* Estimated glomerular filtration rate (Modification of Diet in Renal Disease (MDRD) formula) ≥ 60 ml/min/1.73 m2.

Exclusion Criteria:

* Any significant hepatic, renal, respiratory (e.g., asthma), gastrointestinal, endocrine (e.g., diabetes, dyslipidemia necessitating drug therapy), immunologic, dermatological, hematological, neurologic, psychiatric disease or history of any clinically important drug allergy;
* Acute disease state (e.g., vomiting, fever, diarrhea) within 7 days before study day 1;
* Any history of transient ischemic accident (TIA) or cerebrovascular accident (CVA);
* Any history of acute heart failure or heart failure;
* Any history of myocardial infarction, unstable angina, coronary bypass or percutaneous coronary angioplasty;
* History of malignant tumor during the past 5 years;
* Any medical or surgical disorder considered by the investigator as increasing the risks of participation in the study, or liable to prevent the patient from complying with the requirements of the study or from continuing the study to completion;
* Any situation which, in the investigator's opinion, might compromise assessment of efficacy or of safety;
* History of non-adherence to treatment;
* History of drug abuse within 1 year before study day 1;
* History of alcoholism within 1 year before day 1;
* Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies;
* Use of any investigational drug within 30 days before IMP administration;
* Donation of blood (i.e., 500 ml) within 90 days before study day 1;
* Known secondary hypertension;
* Grade III hypertension;
* Estimated glomerular filtration rate (MDRD formula) below 60 ml/min/1.73 m2 ;
* Type I diabetes mellitus or uncontrolled type II diabetes mellitus (HbA1C ≥ 8%);
* Severe obesity (BMI ≥ 40 kg/m2);
* Arm circumference ≥ 42 cm;
* Atrial fibrillation;
* Known hypersensitivity to drugs;
* History of spontaneous or drug induced angioneurotic edema;
* Use of any of the following medications within the four (4) weeks prior to dosing:

  * Thyroid medication, statin therapy, oral antidiabetic drugs, estrogen replacement therapy and/or chronic low dose aspirin (75 mg/day) unless the patient has been on a stable maintenance dose for at least 3 months prior to screening.
  * Anticoagulant treatments
  * Cholestyramine resins.
  * Treatment with oral, topical, inhaled, eye drop corticosteroids
  * Treatment with class Ia, Ib and Ic or III anti-arrhythmics
  * CNS drugs
  * P-glycoprotein (P-gp) inhibitors (e.g., verapamil, quinidine, ritonavir),
  * known cytochrome P450 inducers or inhibitors (eg, ketoconazole/CYP3A4, quinidine/CYP2D6, gemfibrozil/CYP2C8)
  * Chronic use of nonsteroidal anti-inflammatory drugs (NSAIDS) or cyclooxygenase (COX)-2 inhibitors.
  * Vasodilators or vascular muscle relaxants prescribed for other conditions
* Unlikely to cooperate in the study and/or poor compliance anticipated by the investigator, e.g., uncooperative attitude, inability to return for follow-up visit, and unlikelihood of completing the study;
* Participation in another interventional study at the same time or within 3 months prior to the beginning of the present study;
* Participant not affiliated with the French social security;
* No written informed consent;
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
* A history of additional risk factors for Torsade de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);
* The use of concomitant medications that prolong the QT/QTc interval.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Efficacy - 24h ABPM | Change from Period 1 to Period 2 up to 16 weeks (end-of-study visit).
  Measurements will include mean 24h systolic and diastolic pressures, and daytime values (measured every 15 min from 07:00 am to 10:00 pm) and night-time values (measured every 20 min from 10:00 pm to 07:00 am). Only ambulatory BP recordings with a minimum of 24 measurements will be considered as successful.

SECONDARY OUTCOMES:
Efficacy - Self BP measurements at home | Change from Period 1 to Period 2 up to 16 weeks.
  Additional information will be obtained from self-measurement of BP at home (HBP) with an automatic validated device. To be performed for 7 consecutive days just before the planned visit.
Efficacy - Office BP measurements | Change from Period 1 to Period 2 up to 16 weeks.
  Office SBP, DBP and HR measured after resting in the semi-recumbent position for at least 5 min. Office SBP, DBP and HR measured after 1 min in a standing position will be recorded at each visit, immediately before the administration of the study drug.
Efficacy - Hormonal measurements | Change from Period 1 to Period 2 up to 16 weeks.
  The pharmacodynamic neurohormonal effects of QGC001 will be assessed by measurements of plasma active renin, aldosterone, cortisol, adrenocorticotropic hormone (ACTH), apelin and copeptin as well as urine aldosterone, cortisol, creatinine, sodium and potassium using commercially available validated assays.
Pharmacokinetics - Plasma levels of QGC001 | Change from Period 1 to Period 2 up to 16 weeks.
  Four (4) PK blood samples will be taken. Plasma levels of QGC001 and its metabolite EC33 will be measured using validated LC/MS/MS methods.
Pharmacokinetics - Plasma levels of EC33 | Change from Period 1 to Period 2 up to 16 weeks.
  Four (4) PK blood samples will be taken. Plasma levels of QGC001 and its metabolite EC33 will be measured using validated LC/MS/MS methods.
Safety - Reported signs and symptoms | Change from Period 1 to Period 2 up to 16 weeks.
  Patients will report to the center at approximately 08:00 am, without having taken their morning dose, to undergo safety assessments.
Safety - Physical examination | Change from Period 1 to Period 2 up to 16 weeks.
  The physical examinations will be performed by the investigator or his/her representatives.
Safety - Vital sign measurements | Change from Period 1 to Period 2 up to 16 weeks.
  For OBP measurements, three consecutive (2 min interval) SBP/DBP measurements will be done with an adapted cuff after resting in the semi-recumbent position for at least 5 min using a validated oscillometric semi-automatic device. In addition, SBP, DBP and HR will be measured after 1 min in a standing position.
Safety - Adverse events | Change from Period 1 to Period 2 up to 16 weeks.
Safety - Morisky Medication Adherence Questionnaire | Change from Period 1 to Period 2 up to 16 weeks.
Safety - Electrocardiogram | Change from Period 1 to Period 2 up to 16 weeks.
  The measurements will consist of a 12-lead digital ECG.
Safety - Clinical laboratory tests | Change from Period 1 to Period 2 up to 16 weeks.
  These include blood cells count, fasting glucose, sodium, potassium, chlorides, bicarbonates, creatinine, uric acid, total proteins, total cholesterol, high density lipoprotein (HDL) cholesterol, triglycerides, aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), bilirubin, gamma glutamyl transferase (GammaGT), alkaline phosphatases.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Arthur Gardiner, Dinard
  - Hôpital Cardiologique, CHRU de Lille, Lille
  - Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon
  - Hôpital Européen Georges Pompidou, Paris

REFERENCES:
- [Derived] Khosla J, Aronow WS, Frishman WH. Firibastat: An Oral First-in-Class Brain Aminopeptidase A Inhibitor for Systemic Hypertension. Cardiol Rev. 2022 Jan-Feb 01;30(1):50-55. doi: 10.1097/CRD.0000000000000360. PMID 33027067
- [Derived] Azizi M, Courand PY, Denolle T, Delsart P, Zhygalina V, Amar L, Lantelme P, Mounier-Vehier C, De Mota N, Balavoine F, Llorens-Cortes C. A pilot double-blind randomized placebo-controlled crossover pharmacodynamic study of the centrally active aminopeptidase A inhibitor, firibastat, in hypertension. J Hypertens. 2019 Aug;37(8):1722-1728. doi: 10.1097/HJH.0000000000002092. PMID 30882604